CLINICAL TRIAL: NCT06026540
Title: The Effect of Peer-Guided Pilates Exercise on Premenstrual Syndrome Symptoms and Healthy Lifestyle Behaviors: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/01
Record Dates: First submitted 2023-07-11; First posted 2023-09-07 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-12

CONDITIONS: Premenstrual Syndrome
Keywords: healthy living; Peer guidance; pilates exercise; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After the first measurements were made and the groups were determined; Students in the experimental group will be given pilates exercises 2 days a week for 6 months. Pilates mat, pilates circle, tiny pilates ball and pilates band will be used during the pilates exercise. The duration of the Pilates exercise is 30 minutes in total, and the peer-guided application via "Zoom" includes the following order:
  "Stretching 5 minutes, superman 1 minute, quodratus stretch 2 minutes, marble 1 minute, half plank kick 4 minutes, side kick 4 minutes, pelvic curl 2 minutes, cat pose 1 minute, spine stretch 2 minutes, one leg circle 3 minutes, side leg lift 3 minutes, single leg kick 2 minutes".
  Interventions: Behavioral: Pilates Exercise
- Control group (No Intervention): No intervention will be applied to the control group

INTERVENTIONS:
Behavioral: Pilates Exercise — After the first measurements were made and the groups were determined; Students in the experimental group will be given pilates exercises 2 days a week for 6 months. Pilates mat, pilates circle, tiny pilates ball and pilates band will be used during the pilates exercise. The duration of the Pilates exercise is 30 minutes in total, and the peer-guided application via "Zoom" includes the following order:
  "Stretching 5 minutes, superman 1 minute, quodratus stretch 2 minutes, marble 1 minute, half plank kick 4 minutes, side kick 4 minutes, pelvic curl 2 minutes, cat pose 1 minute, spine stretch 2 minutes, one leg circle 3 minutes, side leg lift 3 minutes, single leg kick 2 minutes".
  Arms: experimental group

SUMMARY:
This project is to examine the effect of pilates exercise, which is applied by university students under the guidance of peers, on premenstrual syndrome symptoms and healthy lifestyle behaviors.

Methods: The research to be carried out within the scope of the project is randomized controlled and has an experimental research design. The population of the research consists of 385 female students studying at the Department of Midwifery at Istanbul University-Cerrahpaşa Faculty of Health Sciences. In the study, it is aimed to reach all students without making a sample calculation in order to identify the students with PMS symptoms among all students. Students who score 110 and above on the Premenstrual Syndrome Scale (PMSS) will be considered to have PMS symptoms. The sample size of the students showing PMS symptoms was determined by using the G*Power (3.1.9.2) program and considering the 0.05 margin of error and data loss, according to 95% power and medium effect size; 27 people should be included in the experimental group and 27 people in the control group. In determining the groups, the participants will be assigned to the experimental and control groups using the "Randomizer.org" program. Students included in the research will be given information about the study and will be presented with an "Informed Consent Form" and a "Volunteer Consent Form". While the experimental group will be given pilates exercises, under the guidance of a peer, for half an hour twice a week for six months, the control group will maintain their routine habits. At the beginning of the study, data will be collected with the "Personal Information Form", "Premenstrual Syndrome Scale (PMSÖ)" and "Healthy Lifestyle Behaviors Scale-II (SYBDS-II)". In the third and sixth months of the study, the hypotheses will be tested by applying PMSS and HLBS-II. The data obtained in the research will be entered into the database in the IBM SPSS 25.0 (Statistical Package for the Social Sciences) program and all necessary statistical analyzes will be performed in the same program.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student studying in the midwifery department of Istanbul University-Cerrahpaşa Faculty of Health Sciences,
* Having a score of 110 and above in PMSS,
* Having an internet connection,
* The Zoom program is installed and ready to use on its electronic device (phone or computer),
* Having the environment to do Pilates.

Exclusion Criteria:

* Being under the age of 18,
* Changes in menstruation characteristics after the diagnosis of PMS,
* Having a chronic or physical illness that prevents Pilates exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Premenstrual Syndrome Scale | 6 months
  The lowest 44 and the highest 220 points can be obtained from the scale. The higher the score, the more severe the PMS problems are. If the person exceeds 50% of the total scale score (110 points in total) on the PMS scale, PMS is considered to be present.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Uncu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Itriyeva K. Premenstrual syndrome and premenstrual dysphoric disorder in adolescents. Curr Probl Pediatr Adolesc Health Care. 2022 May;52(5):101187. doi: 10.1016/j.cppeds.2022.101187. Epub 2022 May 6. PMID 35534402
- [Background] Pearce E, Jolly K, Jones LL, Matthewman G, Zanganeh M, Daley A. Exercise for premenstrual syndrome: a systematic review and meta-analysis of randomised controlled trials. BJGP Open. 2020 Aug 25;4(3):bjgpopen20X101032. doi: 10.3399/bjgpopen20X101032. Print 2020 Aug. PMID 32522750
- [Background] Erbil N, Yucesoy H. Premenstrual syndrome prevalence in Turkey: a systematic review and meta-analysis. Psychol Health Med. 2023 Jun;28(5):1347-1357. doi: 10.1080/13548506.2021.2013509. Epub 2021 Dec 8. PMID 34879766
- [Background] Batibay S, Kulcu DG, Kaleoglu O, Mesci N. Effect of Pilates mat exercise and home exercise programs on pain, functional level, and core muscle thickness in women with chronic low back pain. J Orthop Sci. 2021 Nov;26(6):979-985. doi: 10.1016/j.jos.2020.10.026. Epub 2020 Dec 29. PMID 33386201
- [Background] Tsai SY, Kuo FC, Kuo HC, Liao LL. The prevalence of self-reported premenstrual symptoms and evaluation of regular exercise with premenstrual symptoms among female employees in Taiwan. Women Health. 2018 Mar;58(3):247-259. doi: 10.1080/03630242.2017.1296056. Epub 2017 Mar 20. PMID 28318414